CLINICAL TRIAL: NCT04234789
Title: Predictors of Physical Activity Performance and Dynamic Hyperinflation in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SDC 4245/15/072; 2015/14638-2 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2020-01-08; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Bronchiectasis Adult
Keywords: dynamic hyperinflation; oscillometry; pletysmography
MeSH Terms: interventions — Exercise Test; Spirometry

STUDY DESIGN:
Intervention Model Description: Cross-sectional study. All patients underwent to diagnostic tests protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiopulmonary exercising test (Other): All patients underwent to diagnostic tests protocol
  Interventions: Diagnostic Test: cardiopulmonary exercise testing with dynamic hyperinflation maneuver; Diagnostic Test: spirometry; Diagnostic Test: pletysmography; Diagnostic Test: forced oscillometry technique

INTERVENTIONS:
Diagnostic Test: cardiopulmonary exercise testing with dynamic hyperinflation maneuver — test performed as recommended by ATS guidelines
Diagnostic Test: spirometry — test performed as recommended by ATS guidelines
Diagnostic Test: pletysmography — test performed as recommended by ATS guidelines
Diagnostic Test: forced oscillometry technique — test performed as recommended by ATS guidelines

SUMMARY:
Bronchiectasis is characterized by abnormal and irreversible airway dilation and can be caused by a wide variety of diseases, including congenital diseases, mechanical bronchial obstruction, respiratory infections, and immunodeficiencies. It is a chronic condition with varying severity. Although some patients remain stable for years, the natural history of the disease is progressive deterioration of lung function, Regarding pulmonary function in this group of patients, there are several changes. In a study of 304 patients with bronchiectasis, spirometry was performed in 274 patients. Most of these patients (46.7%) had an obstructive ventilatory disorder, a small percentage of patients (8%) had restrictive disorder and a portion of patients (23.7%) had mixed disorder. The remaining patients (21.5%) had normal spirometry. Dyspnea in this situation occurs due to neuromechanical dissociation, that is, the respiratory drive is increased, but the inspiratory muscles show a reduction in their ability to produce effective ventilation. Besides not knowing if dynamic hyperinflation (DH) is present in patients with bronchiectasis, the mechanism responsible for its onset is also unknown. Exercise capacity is reduced in many patients with bronchiectasis, but there is little information about the exercise response in this population.

The primary objective of this study is to evaluate the prevalence of dynamic hyperinflation in patients with bronchiectasis

DETAILED DESCRIPTION:
Bronchiectasis is characterized by abnormal and irreversible airway dilation and can be caused by a wide variety of diseases, including congenital diseases, mechanical bronchial obstruction, respiratory infections, and immunodeficiencies.

It is a chronic condition with varying severity. Although some patients remain stable for years, the natural history of the disease is progressive deterioration of lung function, chronic respiratory failure, pulmonary hypertension, and right ventricular failure.

Bronchiectasis is a consequence of injury and remodeling with destruction of structural components of the bronchial wall by inflammation and chronic or recurrent infection.The best-known model of developing bronchiectasis is the hypothesis of Cole's vicious cycle. An environmental insult associated with a genetic predisposition impairs mucociliary transport resulting in persistence of microorganisms in the bronchial tree. The infection causes inflammation resulting in tissue damage and further impairing ciliary motility. This leads to further infection, inflammation and lung damage.The patient with bronchiectasis has a cough, chronic sputum, hemoptysis and progressive dyspnea. The clinical course is marked by recurrent infectious exacerbations and over time the patient develops progressive airway obstruction with functional loss.

Regarding pulmonary function in this group of patients, there are several changes. In a study of 304 patients with bronchiectasis, spirometry was performed in 274 patients. Most of these patients (46.7%) had an obstructive ventilatory disorder, a small percentage of patients (8%) had restrictive disorder and a portion of patients (23.7%) had mixed disorder. The remaining patients (21.5%) had normal spirometry.

Dynamic hyperinflation (DH) is characterized by progressive air trapping, which leads to increased end-expiratory lung volume (equivalent to dynamic functional residual capacity) associated with decreased inspiratory capacity (IC) in situations where ventilation is increased, such as exercise. . Dynamic hyperinflation is one of the mechanisms responsible for dyspnea and reduced exercise tolerance in patients with conditions that lead to expiratory flow limitation, such as asthma and COPD.

Studies evaluating dynamic hyperinflation were performed in chronic obstructive pulmonary disease (COPD) patients, demonstrating that the progressive reduction of IC during the maximal or constant load test, on the treadmill or on the cycle ergometer, or through measurements performed before and after the test. The 6-minute walk showed a good correlation with the degree of dyspnea (including the Borg scale) and lower exercise tolerance . Since the total lung capacity (TLC) does not vary or has little non-significant variation during exercise or after bronchodilation, the reduction in IC reflects increased end-expiratory lung volume (VPFE) . In COPD patients, the prevalence of DH is high, around 80% in patients with an average forced expiratory volume in first second (FEV1) of 37%, according to a 2001 study. Asthmatic patients, even with normal spirometry, stable clinical status and no exercise-induced asthma may present limitation to expiratory flow and dynamic hyperinflation during exertion, justifying the presence of dyspnea and less ability to perform exercises In individuals with expiratory flow limitation, the additional elevation of tidal volume (VT) on exertion is limited because operative lung volumes are progressively closer to TLC, in a higher region of the pressure volume curve, where pulmonary compliance is lower. Secondarily, there is a reduction in inspiratory reserve volume (VRI) and, when this volume approaches 500 ml (critical VRI), dyspnea increases considerably, being referred to as inspiratory difficulty. The increase in minute volume is now determined by increased respiratory rate (RR), which further aggravates the situation due to reduced expiratory time (ET), with less time available for elimination of previously inhaled air volume, causing progressive air trapping and worsening pulmonary hyperinflation, entering a vicious cycle (9,10,13,21). Additionally, this mechanism promotes increased elastic overload on the inspiratory muscles by shortening the fibers, reducing their capacity to generate force, determining increased respiratory work, oxygen consumption and the risk of muscle fatigue, as well as adverse hemodynamic effects . Dyspnea in this situation occurs due to neuromechanical dissociation, that is, the respiratory drive is increased, but the inspiratory muscles show a reduction in their ability to produce effective ventilation.

The most commonly used option for dynamic hyperinflation assessment is the serial measurement of IC during maneuvers that promote hyperventilation, such as by performing an incremental or constant-load stress test on the cycle ergometer or treadmill, performing the 6-minute test..

Besides not knowing if DH is present in patients with bronchiectasis, the mechanism responsible for its onset is also unknown. Exercise capacity is reduced in many patients with bronchiectasis, but there is little information about the exercise response in this population. A study was published in 2009 investigating exercise capacity and possible exercise limiting factors in patients with bilateral bronchiectasis. Approximately 50% of patients had reduced exercise capacity, and this was observed in those who had expiratory flow limitation and reduced FEV1 values. Ventilatory limitation, desaturation, and impaired oxygen transport or utilization appear to be the main factors involved in exercise limitation. However, the sample was very small (15 patients) and no DH evaluation was performed.

There are no studies evaluating the presence of DH in patients with bronchiectasis and there are few studies on the physiology of dyspnea in this population. DH is an important mechanism of exercise limitation in COPD and may explain exercise dyspnea and decreased exercise tolerance in patients with bronchiectasis.

Study hypothesis:

Dynamic hyperinflation is present in patients with bronchiectasis.

Objectives:

1. Primary

   - To evaluate the prevalence of dynamic hyperinflation in patients with bronchiectasis
2. Secondary

   * Evaluate aerobic capacity in a population with bronchiectasis
   * To evaluate predictors of dynamic hyperinflation and aerobic limitation in patients with bronchiectasis. Anthropometric data, clinical, functional and tomographic variables will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age followed at the Bronchiectasis Outpatient Clinic of the Pulmonology Department of the University of São Paulo who meet the following criteria will be included in the study:

* Have a diagnosis of bronchiectasis confirmed by chest CT.
* Sign the free and informed consent form for participation in the study.

Exclusion Criteria:

* Diagnosis of Cystic Fibrosis.
* Asthma diagnosis.
* Diagnosis of COPD.
* Pregnancy
* Inability to perform pulmonary function test.
* Recent treatment (<30 days) of infectious exacerbation with oral corticosteroid or antibiotic.
* Contraindication to exercise tests.
* Exercise limitation not related to lung disease (orthopedic or cardiovascular problems).
* History of pulmonary resection.
* Current smoking or previous smoking load greater than 10 years / pack.
* Patients on prolonged home oxygen therapy.
* Allergic bronchopulmonary aspergillosis.
* Active mycobacteriosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of dynamic hyperinflation during cardiopulmonary exercise testing | Day 1 (single visit)
  During cardiopulmonary exercising testing, patients were asked to perform inspiratory capacity maneuvers every 2 minutes. Dynamic hyperinflation was considered as present when the patient had a reduction of 10% or more of the inspiratory capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Athanazio, MD, PhD, Principal Investigator — Medical Assistant
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No